CLINICAL TRIAL: NCT02354313
Title: A Phase III Multicenter, Randomized Study With Lenalidomide Maintenance vs Observation After Induction Regimen Containing Rituximab Followed by High Dose Chemotherapy and ASCT as First Line Treatment in Adult Patients With Advanced Mantle Cell Lymphoma
Brief Title: Phase III, Randomized Trial: Lenalidomide vs Observation After Induction With Rituximab Followed by Cht and ASCT in MCL Adult Patients
Acronym: MCL0208
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIL-MCL0208; 2009-012807-25 (EudraCT Number)
Record Dates: First submitted 2011-06-23; First posted 2015-02-03 (Estimated); Last update posted 2018-02-09 (Actual); Status verified 2018-02

CONDITIONS: MANTLE CELL LYMPHOMA
Keywords: MANTLE CELL LYMPHOMA (MCL); Lenalidomide (Len); Rituximab; ASCT; Revlimid; High dose chemotherapy; transplant
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lenalidomide (Experimental): lenalidomide 10-15 mg once daily on days 1-21, every 28 day, for two years
  Interventions: Drug: Lenalidomide
- Observation (No Intervention): no therapy is planned but only observation

INTERVENTIONS:
Drug: Lenalidomide — Treatment Phase: consisting in an induction phase (3 cycles of RCHOP, given every 21 days); consolidation phase: (high-dose cyclophosphamide (CTX), 2 cycles of high dose Ara-C, BEAM and ASCT).
  Randomization and maintenance phase: Patients who have achieved complete or partial response will be randomized between maintenance with lenalidomide or observation.
  Other Names: Revlimid
  Arms: Lenalidomide

SUMMARY:
A phase III multicenter, randomized study with Lenalidomide (Revlimid®) maintenance versus observation after intensified induction regimen containing rituximab followed by high dose chemotherapy and Autologous Stem Cell Transplantation as first line treatment in adult patients with advanced Mantle Cell Lymphoma: IIL study (MCL0208).

DETAILED DESCRIPTION:
This is a Phase 3, multicenter, open-label, randomized, controlled study to determine the efficacy and safety of lenalidomide as maintenance therapy versus observation in patients with MCL in complete or partial remission after first line intensified and high-dose chemotherapy additioned with rituximab and followed by ASCT. This study will be conducted in three phases: a Screening Phase, a Treatment Phase and a Follow-up Phase

ELIGIBILITY:
Inclusion Criteria.

1. Any male or female adult with newly diagnosed mantle cell lymphoma according to the WHO criteria.
2. Biopsy-proven mantle cell non-Hodgkin's lymphoma, including evidence of cyclin D1 overexpression or the translocation t(11;14)(q13;q32) by FISH or RT-PCR. In subjects whose tumors are negative for the cyclin D1, evidence of overexpression of cyclin D2 or D3 by immunohistochemistry will be acceptable.
3. Age ≥18 years and < 60 with ECOG performance status 0-3, or an age from 60 to 65 years with an ECOG performance status 0-2, except when PS impairment is related to NHL.
4. Advanced stage (Stage III and IV according to Ann Arbor and stage II with bulky disease defined as a mass ≥ 5 cm or B symptoms).
5. Measurable disease (two diameters) in at least one site. Osteoblastic bone lesions, ascites and pleural effusion are not considered measurable disease.
6. Written informed consent prior to any study specific screening procedures, with the understanding that the patient has the right to withdraw from the study at any time, without prejudice.
7. Be willing and able to comply with the protocol for the duration of the study.
8. Females of childbearing potential (FCBP) must: have two negative medically supervised pregnancy test prior to starting of study therapy. She must agree to ongoing pregnancy testing during the course of the study, and after end of study therapy. This applies even if the patient practices complete and continued sexual abstinence. Either commit to continued abstinence from heterosexual intercourse (which must be reviewed on a monthly basis) or agree to use, and be able to comply with, effective contraception without interruption, 28 days prior to starting study drug, during the study therapy (including dose interruptions), and for 28 days after discontinuation of study therapy. The following are effective methods of contraception

   * Implant
   * Levonorgestrel-releasing intrauterine system (IUS)
   * Medroxyprogesterone acetate depot
   * Tubal sterilisation
   * Sexual intercourse with a vasectomised male partner only; vasectomy must be confirmed by two negative semen analyses
   * Ovulation inhibitory progesterone-only pills (i.e., desogestrel)
9. Male patients must agree to use a condom during sexual contact with a FCBP, even if they have had a vasectomy, throughout study drug therapy, during any dose interruption and after cessation of study therapy. Agree to not donate semen during study drug therapy and for a period after end of study drug therapy.
10. All patients must have an understanding that the study drug could have a potential teratogenic risk. They must agree to abstain from donating blood while taking study drug therapy and following discontinuation of study drug therapy. They must to agree not to share study medication with another person. They must be counseled about pregnancy precautions and risks of fetal exposure.

Exclusion Criteria:

1. Non-Hodgkin's lymphoma subtypes other than MCL
2. Cytological variant with small cells with round nuclei mimicking CLL, which is frequently recognized in patients with a leukemic and splenomegaly presentation without or with minimal involvement of lymph nodes and has an indolent clinical course.
3. History of malignancy other than squamous cell carcinoma, basal cell carcinoma of the skin or carcinoma in situ of the cervix, carcinoma in situ of the breast, incidental histological finding of prostate cancer (TNM stage of T1a or T1b) within the last 3 years.
4. Major surgery, other than diagnostic surgery, within the last 4 weeks.
5. Evidence of CNS involvement, patients with an history of uncontrolled seizures, central nervous system disorders or psychiatric disability considered by the Investigator to be clinically significant and adversely affecting compliance to study drugs. If clinically indicated, lumbar puncture, and MRI should be performed during the screening process.
6. Clinically significant cardiac disease (VEF <45%) (e.g. congestive heart failure, symptomatic coronary artery disease and cardiac arrhythmias not well controlled with medication) or myocardial infarction within the last 6 months (New York Heart Association Class III or IV heart disease) and marked impairment of pulmonary function (pulmonary diffusing capacity <50%).
7. Unacceptable hematologic values in the week prior to the start of study: hemoglobin <9 g/dL, WBC <3x109/L, platelets <60x109/L, absolute neutrophil count (ANC)<1.5x109/L (unless cytopenia is secondary to bone marrow involvement or autoimmune cytopenia related to lymphoma).
8. Abnormal liver function tests, within one week prior to study start above any of the values listed: serum bilirubin > 2 mg/dL, ALT or AST >3 times the upper normal value; alkaline phosphatase>2.5 times the upper normal value (unless these abnormalities are due to liver involvement of lymphoma).
9. Abnormal renal function (serum creatinine >2.0 mg/dL), unless it is disease related
10. Patients with active opportunistic infections.
11. Known seropositive for or active viral infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV). Patients who are seropositive because of hepatitis B virus vaccine are eligible. Patients with HBcAb serology, will not be excluded from the study and be given lamivudine as prophylaxis starting one week before chemotherapy. HbsAg and AST/ALT ifHBV DNA is not available, will be monitored every three weeks. If HBV DNA is available, it will be monitored along with HBsAg
12. Pregnant or lactating females

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2010-05 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | 30 months from randomisation
  PFS will be defined as the time between the date of randomization and the date of disease progression, relapse or death from any cause.therapy to prolong progression-free survival (PFS) after completion of first-line high-dose chemotherapy additioned with rituximab and followed by ASCT in adult patients with MCL who have achieved complete response (CR) or partial response (PR). PFS is defined according to Cheson et al (JCO, 2007) as the time from randomisation until lymphoma progression or death as a result of any cause.

SECONDARY OUTCOMES:
Overall Survival (OS) | 36 months from randomisation (42 months from accrual)
  OS will be defined as the time between the date of randomization and the date of death from any cause
Progression Free Survival (PFS) | 36 months from accrual
  PFS will be defined as the time between the date of enrolment and the date of disease progression, relapse or death from any cause.
Disease-free survival (DFS) | 30 months from randomisation (36 months from accrual)
  DFS will be defined in CR patients as the time between the date of randomization and the date of relapse or death as a result of lymphoma or acute toxicity of treatment according to the Cheson 2007
Event-free survival (EFS) | 30 months from randomisation (36 months from accrual)
  EFS will be defined in CR patients as the time between the date of randomization and the date of failure of treatment or death as a result of any cause according to the Cheson 2007
Complete Response (CR) Rate | up to 3 months from accrual
  Proportion of CR according to the Cheson 2007 response criteria
Overall Response Rate (ORR) | up to 3 months from accrual
  ORR is defined as Complete Response (CR) or Partial Response (PR) according to the Cheson 2007 response criteria
Incidence of grade 3 or higher Toxicity measured by CTCAE v.4 at any time during therapy and follow-up. | 30 months from accrual
  Toxicity amount of grade 3 or more as CTCAE
Quality of life | baseline, 6-12-18-24 months from randomisation
  EORTC QLQC30 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Cortelazzo, MD, Study Director — Humanitas Gavazzeni - Bergamo, Lombardia
Locations (53):
- Italy (52):
  - UO Ematologia Ospedale Dell'Angelo, Mestre, VE
  - SC Ematologia A.O.SS. Biagio e Antonio e C. Arrigo, Alessandria
  - AORN San G.Moscati, Avellino
  - Centro di riferimento Oncologico - Oncologia Medica A, Aviano (PN)
  - Istituto di Ematologia ed Oncologia Medica A. Seragnoli Policlinico S. Orsola, Bologna
  - Divisione di Ematologia e TMO, Ospedale di Bolzano, Bolzano
  - Divisione di Ematologia Spedali Civili, Brescia
  - Divisione di Ematologia Osp.Businco, Cagliari
  - IRCC Onco-Ematologia, Candiolo
  - S.C. di Ematologia e Trapianto di Midollo Osseo ASO S. Croce e Carle, Cuneo
  - Divisione di Ematologia, Policlinico Careggi, Florence
  - Ematologia, A.O.U. San Martino, Genova
  - Clinica Ematologica, A.O.U. San Martino - IST, Genova
  - Divisione di Ematologia Ospedale Vito Fazzi, Lecce
  - Istituto Scientifico Romagnolo per lo studio e la cura dei Tumori-IRST - Meldola / Cesena, Meldola (FC)
  - Ematologia AO Ospedali Riuniti Papardo-Piemonte, Messina
  - Divisione di Ematologia, Ospedale Niguarda, Milan
  - Dipartimento di Ematologia e Oncologia - Ospedale Maggiore Policlinico Mangiagalli e Regina Elena, Milan
  - Unità Linfomi- Dipartimento Oncoematologia- Istituto Scientifico San Raffaele IRCCS, Milan
  - Dipartimento di Scienze Mediche UOC di Oncologia ed Ematologia Oncologica - Ospedale di Mirano, Mirano
  - Dip. di Oncologia ed Ematologia - Università di Modena e Reggio Emilia Policlinico - COM Centro Oncologico Modenese, Modena
  - Osp.San Gerardo Divisione di Ematologia, Monza
  - S.C.D.U Ematologia Azienda Ospedaliera Universitaria Maggiore - Università del Piemonte Orientale, Novara
  - U.O.C. Ematologia e CTMO Presidio Ospedale S. Francesco, Nuoro
  - U.O. Oncoematologia Ospedale "Andrea Tortora", Pagani
  - Divisione di Ematologia, Azienda Ospedali Riuniti Villa Sofia Cervello, Palermo
  - Oncoematologia e TMO Clinica "La Maddalena", Palermo
  - Cattedra di Ematologia - Centro Trapianti Midollo Osseo - Università Parma, Parma
  - Fondazione Policlinico San Matteo Clinica Ematologica, Pavia
  - U.O. Ematologia e Centro Trapianto Midollo Osseo - Ospedale G. da Saliceto, Piacenza
  - Dipartimento di Oncologia Divisione di Ematologia, Azienda Ospedaliera Pisana Ospedale "S.Chiara", Pisa
  - Divisione di Ematologia con TMO - Ospedale San Carlo, Potenza
  - U.O di Ematologia Ospedale S. Maria delle Croci, Ravenna
  - Divisione di Ematologia - Presidio Ospedali Riuniti Bianchi, Melacrino, Morelli, Reggio Calabria
  - S. C. Ematologia - Azienda Ospedaliera Arcispedale - "S.Maria Nuova" IRCCS, Reggio Emilia
  - UO Ematologia - Ospedale degli Infermi, Rimini
  - Cattedra di Ematologia Università Cattolica Policlinico Gemelli, Roma
  - Dipartimento di Biotecnologie Cellulari ed Ematologia Università "La Sapienza", Roma
  - Divisione di Ematologia Policlinico Università Tor-Vergata, Roma
  - Divisione di Oncologia Medica ed Ematologia, Istituto Clinico Humanitas, Rozzano (MI)
  - Divisione di Ematologia, Centro Trapianto di Cellule Staminali, IRCCS "Casa Sollievo della Sofferenza", San Giovanni Rotondo
  - Istituto di Ematologia - Azienda Ospedaliero Universitaria di Sassari, Sassari
  - Divisione di Ematologia - Policlinico Le Scotte, Siena
  - Struttura Complessa di Oncoematologia - Ospedale Santa Maria, Terni
  - S.C.D.U. Ematologia Universitaria A.O. Città della Salute e della Scienza di Torino, Torino
  - SC. Ematologia A.O. Città della Salute e della Scienza, Torino
  - Divisione di Ematologia ASL BAT 1, Trani
  - U.O. Ematologia e Immunoematologia - Ospedale Cà Foncello, Treviso
  - Divisione di Ematologia Ospedale Cardinale Panico, Tricase
  - Ematologia Clinica Ospedale Maggiore, Trieste
  - Clinica Ematologica ASUI Integrata di Udine, Udine
  - Ospedale Policlinico G.B. Rossi, Verona
- Departemento de Hematologia di Instituto Português de Oncologia de Lisboa Francisco Gentil, Lisbon, Portugal

REFERENCES:
- [Derived] Ragaini S, Galli A, Genuardi E, Gandossini M, Alessandria B, Civita AM, Evangelista A, Amaducci E, Stefoni V, Cavallo F, Ballerini F, Puccini B, Vallisa D, Michieli M, Pascarella A, Palmas A, Patti C, Lucchini E, Careddu MG, Merli M, Postorino M, Boccomini C, Balzarotti M, Zilioli VR, Gomes da Silva M, Bruno B, Rizzo E, Ladetto M, Malcovati L, Ferrero S. Large clones of clonal hematopoiesis affect outcome in mantle cell lymphoma: results from the FIL MCL0208 clinical trial. Blood Adv. 2025 Apr 22;9(8):1805-1815. doi: 10.1182/bloodadvances.2024014948. PMID 39808795
- [Derived] Zaccaria GM, Ferrero S, Hoster E, Passera R, Evangelista A, Genuardi E, Drandi D, Ghislieri M, Barbero D, Del Giudice I, Tani M, Moia R, Volpetti S, Cabras MG, Di Renzo N, Merli F, Vallisa D, Spina M, Pascarella A, Latte G, Patti C, Fabbri A, Guarini A, Vitolo U, Hermine O, Kluin-Nelemans HC, Cortelazzo S, Dreyling M, Ladetto M. A Clinical Prognostic Model Based on Machine Learning from the Fondazione Italiana Linfomi (FIL) MCL0208 Phase III Trial. Cancers (Basel). 2021 Dec 31;14(1):188. doi: 10.3390/cancers14010188. PMID 35008361
- [Derived] Ladetto M, Cortelazzo S, Ferrero S, Evangelista A, Mian M, Tavarozzi R, Zanni M, Cavallo F, Di Rocco A, Stefoni V, Pagani C, Re A, Chiappella A, Balzarotti M, Zilioli VR, Gomes da Silva M, Arcaini L, Molinari AL, Ballerini F, Ferreri AJM, Puccini B, Benedetti F, Stefani PM, Narni F, Casaroli I, Stelitano C, Ciccone G, Vitolo U, Martelli M. Lenalidomide maintenance after autologous haematopoietic stem-cell transplantation in mantle cell lymphoma: results of a Fondazione Italiana Linfomi (FIL) multicentre, randomised, phase 3 trial. Lancet Haematol. 2021 Jan;8(1):e34-e44. doi: 10.1016/S2352-3026(20)30358-6. Epub 2020 Dec 22. PMID 33357480
- [Derived] Zaccaria GM, Ferrero S, Rosati S, Ghislieri M, Genuardi E, Evangelista A, Sandrone R, Castagneri C, Barbero D, Lo Schirico M, Arcaini L, Molinari AL, Ballerini F, Ferreri A, Omede P, Zamo A, Balestra G, Boccadoro M, Cortelazzo S, Ladetto M. Applying Data Warehousing to a Phase III Clinical Trial From the Fondazione Italiana Linfomi Ensures Superior Data Quality and Improved Assessment of Clinical Outcomes. JCO Clin Cancer Inform. 2019 Oct;3:1-15. doi: 10.1200/CCI.19.00049. PMID 31633999
- [Derived] Ferrero S, Rossi D, Rinaldi A, Bruscaggin A, Spina V, Eskelund CW, Evangelista A, Moia R, Kwee I, Dahl C, Di Rocco A, Stefoni V, Diop F, Favini C, Ghione P, Mahmoud AM, Schipani M, Kolstad A, Barbero D, Novero D, Paulli M, Zamo A, Jerkeman M, da Silva MG, Santoro A, Molinari A, Ferreri A, Gronbaek K, Piccin A, Cortelazzo S, Bertoni F, Ladetto M, Gaidano G. KMT2D mutations and TP53 disruptions are poor prognostic biomarkers in mantle cell lymphoma receiving high-dose therapy: a FIL study. Haematologica. 2020 Jun;105(6):1604-1612. doi: 10.3324/haematol.2018.214056. Epub 2019 Sep 19. PMID 31537689
- [Derived] Bomben R, Ferrero S, D'Agaro T, Dal Bo M, Re A, Evangelista A, Carella AM, Zamo A, Vitolo U, Omede P, Rusconi C, Arcaini L, Rigacci L, Luminari S, Piccin A, Liu D, Wiestner A, Gaidano G, Cortelazzo S, Ladetto M, Gattei V. A B-cell receptor-related gene signature predicts survival in mantle cell lymphoma: results from the Fondazione Italiana Linfomi MCL-0208 trial. Haematologica. 2018 May;103(5):849-856. doi: 10.3324/haematol.2017.184325. Epub 2018 Feb 22. PMID 29472356